CLINICAL TRIAL: NCT02938221
Title: Feasibility and Safety of a Telemedically Performed Three-Component Oculomotor Testing Battery (HINTS) in Healthy Adults
Brief Title: Telemedical Examination of a Three-Component Oculomotor Testing Battery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Munich Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TeleHINTS-1
Record Dates: First submitted 2016-10-14; First posted 2016-10-19 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Stroke; Vertigo; Dizziness
Keywords: TeleStroke; HINTS; Diagnosis; Telemedicine; Acute Vestibular Syndrome
MeSH Terms: conditions — Stroke; Vertigo; Dizziness; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telemedical video-oculography (Experimental): Execution of three oculomotor tests using a telemedical video-oculography system
  Interventions: Device: Telemedical video-oculography system

INTERVENTIONS:
Device: Telemedical video-oculography system — Telemedical video-oculography setup consisting of video goggles (EyeSeeCam, Interacoustics GmbH, Germany), a mobile telemedical workstation and an extended conferencing and remote control system (MEYTEC GmbH, Germany)

SUMMARY:
The study investigates the feasibility and safety of the telemedical implementation of three diagnostic oculomotor tests using a video-oculography device and an extended teleconferencing system. The testing battery comprises Halmagyi's head impulse test, test for nystagmus and test of skew (vertical misalignment) known as the HINTS protocol. Previously published data have shown high sensitivity and specificity of the protocol for the discrimination of central and peripheral causes of acute vestibular syndrome. In this study the three tests will be executed on 30 healthy subjects using video goggles (EyeSeeCam, Interacoustics GmbH, Germany) connected to a mobile wireless-workstation for bidirectional audiovisual communication in a clinical environment (MEYTEC GmbH, Germany). A newly developed remote control and video conferencing solution allows the execution and evaluation of the HINTS protocol in a telemedical setup.

The examination is guided by a remote physician using the help of a trained assistant attending to the subject. Corresponding clinical bedside tests will be executed for comparison. Primary endpoint is feasibility of the three diagnostic tests in a telemedical setting. Safety as well as accuracy of the telemedical versus bedside examination will be analyzed as secondary outcome measures. Aim of the study is to improve diagnostic accuracy for patients with acute vestibular syndrome in remote areas where specialists are rare.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults

Exclusion Criteria:

* Acute vertigo or dizziness, acute neck pain, history of stroke, history of acute vestibular syndrome, strong unilateral or bilateral visual impairment, complete movement restriction of cervical spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of evaluable telemedical oculomotor examinations | through completion of diagnostic test, an average of 10 minutes

SECONDARY OUTCOMES:
Accuracy of telemedical oculomotor examination (correlation to bedside test) | through completion of diagnostic test, an average of 10 minutes
Number of participants with adverse or serious adverse events that are related to telemedical oculomotor examination | through completion of diagnostic test, an average of 10 minutes
Time delay of telemedical tests | through completion of diagnostic test, an average of 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gordian J Hubert, Dr. med., Principal Investigator — Städtisches Klinikum München GmbH
Locations (1):
- Klinikum München-Harlaching, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kattah JC, Talkad AV, Wang DZ, Hsieh YH, Newman-Toker DE. HINTS to diagnose stroke in the acute vestibular syndrome: three-step bedside oculomotor examination more sensitive than early MRI diffusion-weighted imaging. Stroke. 2009 Nov;40(11):3504-10. doi: 10.1161/STROKEAHA.109.551234. Epub 2009 Sep 17. PMID 19762709
- [Background] Newman-Toker DE, Kerber KA, Hsieh YH, Pula JH, Omron R, Saber Tehrani AS, Mantokoudis G, Hanley DF, Zee DS, Kattah JC. HINTS outperforms ABCD2 to screen for stroke in acute continuous vertigo and dizziness. Acad Emerg Med. 2013 Oct;20(10):986-96. doi: 10.1111/acem.12223. PMID 24127701
- [Background] Bartl K, Lehnen N, Kohlbecher S, Schneider E. Head impulse testing using video-oculography. Ann N Y Acad Sci. 2009 May;1164:331-3. doi: 10.1111/j.1749-6632.2009.03850.x. PMID 19645921
- [Background] MacDougall HG, Weber KP, McGarvie LA, Halmagyi GM, Curthoys IS. The video head impulse test: diagnostic accuracy in peripheral vestibulopathy. Neurology. 2009 Oct 6;73(14):1134-41. doi: 10.1212/WNL.0b013e3181bacf85. PMID 19805730
- [Background] Newman-Toker DE, Saber Tehrani AS, Mantokoudis G, Pula JH, Guede CI, Kerber KA, Blitz A, Ying SH, Hsieh YH, Rothman RE, Hanley DF, Zee DS, Kattah JC. Quantitative video-oculography to help diagnose stroke in acute vertigo and dizziness: toward an ECG for the eyes. Stroke. 2013 Apr;44(4):1158-61. doi: 10.1161/STROKEAHA.111.000033. Epub 2013 Mar 5. PMID 23463752